CLINICAL TRIAL: NCT02651779
Title: Internal Plate Fixation vs. Plaster in Complete Articular Distal Radial Fractures
Acronym: VIPAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dijklander Ziekenhuis (Other); Maasstad Hospital (Other); Maxima Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other); Rijnland Hospital (Other); Diakonessenhuis, Utrecht (Other); BovenIJ Hospital (Other); Onze Lieve Vrouwe Gasthuis (Other); Groene Hart Ziekenhuis (Other); Reinier de Graaf Groep (Other); Flevoziekenhuis (Other); Ziekenhuis Rivierenland (Other); Radboud University Medical Center (Other); Ziekenhuis Amstelland (Other); Medical Center Alkmaar (Other); Red Cross Hospital Beverwijk (Other); Zaans Medical Center (Unknown)
Responsible Party: Principal Investigator, J.C. Goslings, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL51544.018.14
Record Dates: First submitted 2016-01-04; First posted 2016-01-11 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Displaced Complete Articular Distal Radius Fractures
MeSH Terms: interventions — Open Fracture Reduction; Surgical Procedures, Operative; POLR1G protein, human; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed reduction and plasterimmobilisation (Active Comparator): The control group will be treated with closed reduction and cast immobilization. This will take place under local anaesthesia by means of a haematoma block with 20 cc Lidocaine 1%. Closed reduction will be preferably performed according to the Robert-Jones method. This involves increasing the deformity first, then applying continuous traction and immobilizing wrist and hand in the reduced position. Additional radiographs will be performed to verify the success of the reduction. After this has been confirmed, the wrist will be immobilized initially in a split plaster and later changed into a circular cast for five to six weeks immobilization in total.
  Interventions: Other: Closed reduction and plasterimmobilisation
- Open reduction and internal plate fixation (Other): The surgery will be performed by a certified trauma surgeon. According to the current standard treatment protocol, antibiotic prophylaxis will be administered thirty minutes preoperatively. The distal radius will be approached according to Henry, which beholds an incision between the tendon of the flexor carpi radialis muscle and the radial artery. After the fracture site is exposed, the fracture will be reduced and provisionally fixed under fluoroscopy with K-Wires/reduction forceps. An appropriate volar locking plate which best suits the anatomy of the wrist and the fracture type will be selected. Fracture reduction and screw placement will be confirmed by radiographic images. Additionally, fixation can be supported by a dorsal plate or radial column plate. This will be at discretion of the surgeon and depends on the fracture configuration and the position of the fragments. Wound closure will be performed at the discretion of the surgeon using standard techniques.
  Interventions: Procedure: Open reduction and internal plate fixation

INTERVENTIONS:
Procedure: Open reduction and internal plate fixation
  Other Names: ORIF; Surgical treatment
  Arms: Open reduction and internal plate fixation
Other: Closed reduction and plasterimmobilisation
  Other Names: Cast; Conservative treatment
  Arms: Closed reduction and plasterimmobilisation

SUMMARY:
There is no consensus about the best treatment for patients with displaced complete articular distal radius fractures (AO type C fractures). Despite this lack of consensus and the lack of available literature on comparative data to guide treatment for this patient population, operative treatment with plate fixation has gained popularity. The aim of this study is to compare the functional outcome of open reduction and plate fixation with closed reduction and plaster immobilisation in adult patients (18-75 years) with displaced complete articular distal radius fractures.

DETAILED DESCRIPTION:
Distal radius fractures account for 17% of all fractures diagnosed. Two third of those fractures are displaced and need to be reduced.

According to the Dutch National Guidelines, displaced distal radius fractures, after adequate reduction confirmed on X-ray, are best treated nonoperatively with cast immobilization. Moreover, the AAOS Clinical Practice Guideline only suggest surgical fixation when the articular step, after reduction, exceeds 2mm. However, both recommendations are based on studies who did not differentiate between intra- and extra-articular distal radius fractures. So, no clear consensus about the best treatment for patients with displaced intra-articular distal radius fractures can be made. Despite this lack of consensus and the lack of available literature on comparative data to guide treatment for this patient population, a rise in use of volar plating has been observed.

The goal of open reduction and plate fixation is to restore articular congruity and axial alignment, and to enable early post-operative movement. Several studies show good radiological and functional results using the volar locking plate in unstable displaced distal radius fractures.

No studies have been carried out to assess whether operative treatment with plate fixation is superior in displaced complete articular distal radius fractures to nonoperative treatment in patients with these fracture type. Therefore, with this randomized controlled trial the investigators wish to determine the difference in functional outcome, assessed with the Patient Related Wrist Evaluation (PRWE), after open reduction and plate fixation compared to nonoperative treatment with closed reduction and cast immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 - 75 years
* AO type C displaced distal radius fracture, as classified on lateral, posterior anterior and lateral carporadial radiographs/CT-scan by a radiologist or trauma surgeon
* Acceptable closed reduction obtained immediately after admission to the Emergency Department (<12hrs)

Exclusion Criteria:

* Patients with impaired wrist function prior to injury due to arthrosis/neurological disorders of the upper limb
* Open distal radius fractures
* Multiple trauma patients (Injury Severity Score (ISS) ≥16)
* Other fractures of the affected extremity (except from ulnar styloid process)
* Fracture of other wrist
* Insufficient comprehension of the Dutch language to understand a rehabilitation program and other treatment information as judged by the attending physician
* Patient suffering from disorders of bone metabolism other than osteoporosis (i.e. Paget's disease, renal osteodystrophy, osteomalacia)
* Patients suffering from connective tissue disease or (joint) hyperflexibility disorders such as Marfan's, Ehler Danlos or other related disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Wrist pain and disability measured with the Patient Rated Wrist Evaluation (PRWE) | 12 months
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living. The PRWE allows patients to rate their levels of wrist pain and disability from 0 to 10, and consists of three subscales: Pain, Function and Cosmetics.

SECONDARY OUTCOMES:
Disability of the wrist measured with the Disability of the Arm, Shoulder and Hand (DASH) questionnaire | 6 weeks and 3, 6 and 12 months
  The Disabilities of the Arm, Shoulder and Hand (DASH) score is a 30-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb.
Quality of life measured with the SF-36 | 6 weeks and 3, 6 and 12 months
  Quality of Life assessed using the Short Form-36 (SF-36) questionnaire. The SF-36 is a validated multipurpose, short form health survey which contains 36 questions representing eight different health domains. These domains are combined into a mental and physical component scale. From each domain, scores ranging from 0 to 100 points are derived, with lower scores indicating poorer quality of life.
Pain measured with the Visual Analogue Scale (VAS) | 1, 3 and 6 weeks and 3, 6 and 12 months
  Pain as indicated on a visual Analogue Scale (VAS), in which 0 implies no pain and 10 the worst possible pain. Patients will be asked to give an estimation of the type and quantity of pain medication taken during all follow-up visits.
Range of motion measured with a goniometer | 6 weeks and 3, 6 and 12 months
  Range of motion of the wrist measured on both sides with a handheld goniometer in degrees. ROM includes pronation and supination, ulnar and radial deviation and palmar and dorsal flexion of the wrist.
Grip strength measured with a dynamometer | 6 weeks and 3, 6 and 12 months
  Grip strength as measured with a dynamometer in kg as the mean of three measurements. Grip strength will be measured as a percentage of the uninjured side.
Number of patients with loss of reduction | 1, 3 and 6 weeks and 3, 6 and 12 months
  Radiographs will be performed to ensure that loss of reduction has not occurred. Loss of reduction is defined as <15° radial inclination, >15° of dorsal angulation or >20° of volar angulation, >3 mm shortening of ulnar variance or >2 mm of articular step-off or gap. Radial inclination, volar/dorsal tilt, ulnar variance and radial length will be measured digitally in the Picture Archiving and Communication System (PACS) on standard posterior anterior (PA), lateral carporadial and lateral X-rays of the wrist. If loss of reduction occured, operative treatment will be considered, but will be at discretion of the treating surgeon.
Cost-effectiveness and cost-utility measured with an economic evaluation questionnaire | 6 weeks and 3, 6 and 12 months
  Cost-effectiveness and cost-utility measured with an economic evaluation questionnaire based on the EQ-6D and the Standard Form Health and Labour questionnaire.
Number of complications in both treatment groups | 1, 3 and 6 weeks and 3, 6 and 12 months
  Number of complications in both patients treated with plasterimmobilisation and ORIF. Complications include loss of reduction, cross-overs from conservative to operative treatment, fracture malunion or non-union, wound and/or plate infection, tendon irritation and/or rupture, neuropathy and the occurrence of complex regional pain syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: J. Carel Goslings, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Niels W.L. Schep, MD, PhD, MSc, Principal Investigator — Maasstad Hospital
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Mulders MAM, Walenkamp MMJ, Goslings JC, Schep NWL. Internal plate fixation versus plaster in displaced complete articular distal radius fractures, a randomised controlled trial. BMC Musculoskelet Disord. 2016 Feb 9;17:68. doi: 10.1186/s12891-016-0925-y. PMID 26860090